CLINICAL TRIAL: NCT07128797
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled Phase Ib Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Subcutaneous Injections of B1344 Injection in Patients With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: a Safety, Tolerability, and Pharmacokinetic Trial of Multiple Subcutaneous Injections of B1344 Injection in Patients With Nonalcoholic Fatty Liver Disease（NAFLD）
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASLY-BM-B1344-NASH-Ib
Record Dates: First submitted 2025-07-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: NAFLD (Non-alcoholic Fatty Liver Disease); NASH (Nonalcoholic Steatohepatitis)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- B1344 30mg weekly (QW) (Experimental)
  Interventions: Drug: B1344
- B1344 45mg weekly (QW) (Experimental)
  Interventions: Drug: B1344
- B1344 60mg Every 2 Weeks (Q2W) (Experimental)
  Interventions: Drug: B1344
- B1344 90mg Every 2 Weeks (Q2W) (Experimental)
  Interventions: Drug: B1344
- Placebo QW or Q2W (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: B1344 — Subcutaneous injection
  Arms: B1344 30mg weekly (QW); B1344 45mg weekly (QW); B1344 60mg Every 2 Weeks (Q2W); B1344 90mg Every 2 Weeks (Q2W)
Other: Placebo — Subcutaneous injection
  Arms: Placebo QW or Q2W

SUMMARY:
This is a randomized, double-blind, multicenter, placebo-controlled, multiple-dose escalating clinical trial designed to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity profile of B1344 in patients with NAFLD. Additionally, the trial will conduct preliminary observations on the efficacy of B1344, aiming to provide early proof of concept for B1344 as a therapeutic agent for NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese patients aged between 18 and 75 years;
2. Patients diagnosed with NAFLD and with a magnetic resonance proton density fat fraction (MRI-PDFF) ≥10% in the screening/baseline period or within one month prior;
3. Presence of any one of the following metabolic risk factors:

   * Body Mass Index (BMI) ≥24.0 kg/m² or abdominal obesity (male waist circumference ≥90 cm, female waist circumference ≥85 cm);
   * Fasting blood glucose ≥6.1 mmol/L, or 2-h blood glucose after glucose load ≥7.8 mmol/L, or glycated hemoglobin (HbA1c) ≥5.7%, or history of type 2 diabetes, or Homeostasis Model Assessment Insulin Resistance Index (HOMA-IR) ≥2.5;
   * Resting blood pressure ≥130/85 mmHg, or currently receiving antihypertensive medication;
   * Fasting serum triglycerides (TG) ≥1.70 mmol/L, high-density lipoprotein cholesterol (HDL-c) ≤1.0 mmol/L (male) and 1.3 mmol/L (female), or currently receiving lipid-lowering medication.
4. Weight stability reported by participants within 6 weeks before enrollment (absolute weight change ≤5%).
5. Participants have no fertility plans within 3 months after signing the informed consent and voluntarily take effective contraceptive measures.
6. Voluntary participation in the clinical trial, able to sign the informed consent, and capable of understanding and complying with the trial procedures.

Exclusion Criteria:

1. Liver biopsy, or clinical diagnosis of cirrhosis based on clinical presentation, biochemical and imaging results, or any of the following criteria: ① FIB-4 score ≥3.48 in the screening/baseline period or within 1 month prior, or liver stiffness value (LSM) ≥15 kPa based on FibroScan; ② liver biopsy results indicating NASH-F4 stage within the previous 24 months; ③ clinical examination signs of liver cirrhosis or splenomegaly during the screening/baseline period; ④ abdominal imaging results showing liver nodules or splenomegaly during the screening/baseline period or within 1 month prior.
2. History of tumors or liver transplantation, or patients planning to undergo liver transplantation.
3. History of liver diseases other than NAFLD or clinical suspicion of liver diseases other than NAFLD, including but not limited to secondary NAFLD, hepatitis B, hepatitis C, autoimmune hepatitis, hemochromatosis, alcoholic liver disease, primary sclerosing cholangitis, primary biliary cholangitis, or Wilson's disease.
4. History of other diabetes besides T2DM (such as type 1 diabetes, secondary diabetes, etc.), or currently using or planning to use insulin, thiazolidinediones, and glucagon-like peptide-1 (GLP-1) analog drugs for treatment.
5. Presence of other severe, progressive, or uncontrolled diseases besides T2DM, hypertension, and dyslipidemia, including but not limited to immune system, endocrine system, hematologic system, urinary system, hepatobiliary system, respiratory system, nervous system, psychiatric system, cardiovascular system, digestive system, where participation in this trial would increase participant risk as determined by the investigator.
6. Previous history of weight-loss surgery or plans for weight-loss during the trial, or significant changes in exercise or dietary habits.
7. History of extra-bone injury, fracture, or bone-related surgery within 2 months before screening.
8. Participants with a history of long QT syndrome or family history of sudden death, or males with QTcF > 450 ms, females with QTcF > 470 ms.
9. Allergic to B1344 or its excipients, or history of allergy to other biological products or severe allergic reactions.
10. History of drug use related to secondary NAFLD lasting more than 2 weeks within 12 months before screening, including amiodarone, methotrexate, systemic corticosteroids, 5-fluorouracil, irinotecan, tetracycline, tamoxifen, doses exceeding hormone replacement estrogen, anabolic steroids, valproic acid, and other known hepatotoxic drugs.
11. History of concomitant treatment that does not meet protocol requirements before enrollment, or concomitant treatment that meets protocol requirements but cannot maintain a stable dose until the end of the trial, or plans to initiate new concomitant treatments after the first dose until the end of the trial.
12. Previous use of FGF-21 analogs or FGFR1 agonists.
13. Screening/baseline examination results meeting the following criteria:

    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥5 times the upper limit of normal (ULN), total bilirubin >ULN;
    * Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m²;
    * Hemoglobin <120 g/L (male) or <110 g/L (female);
    * HbA1c ≥9%; fasting blood glucose ≥13.9 mmol/L;
    * International normalized ratio (INR) >1.3;
    * Platelet count <110×10⁹/L;
    * Dual-energy X-ray absorptiometry (DXA) T-score ≤-2.5;
    * Resting systolic blood pressure <90 or ≥160 mmHg, resting diastolic blood pressure <50 or ≥100 mmHg;
    * Resting heart rate <60 or >100 beats/minute;
    * TG ≥5.65 mmol/L;
    * Hepatitis B surface antigen (HBsAg) positive, hepatitis C antibody (HCVAb) positive, human immunodeficiency virus (HIV) antibody positive, or positive for serum Treponema pallidum specific antibody (TP-Ab).
14. History of long-term excessive alcohol consumption, or alcohol consumption ≥14 World Health Organization (WHO) alcohol units per week (1 WHO alcohol unit = 10 g pure alcohol) within 3 months before screening, or positive alcohol screening, or unable to refrain from alcohol 48 hours before the first dose until the end of the trial.
15. Excessive consumption of tea, coffee, or caffeinated beverages (daily consumption of more than 8 cups of respective drinks, with 1 cup being 250 mL) within 3 months before screening, or consumption of any caffeinated food or drink (such as coffee, strong tea, chocolate, cola, etc.) within 48 hours before the first dose.
16. History of blood donation, loss of blood ≥200 mL, blood transfusion, or use of blood products within 3 months before screening, or plans to donate blood during the trial.
17. History of needle phobia, blood phobia, or frequent episodes of orthostatic hypotension, or inability to tolerate venipuncture.
18. History of drug abuse, or positive urine drug abuse screening.
19. Smoking more than 5 cigarettes daily within the last 3 months or cannot completely quit smoking during the trial.
20. Women who are pregnant or breastfeeding, or planning to become pregnant or breastfeed during the trial.
21. Any skin or abdominal wall anomalies that would affect subcutaneous injection, or tattoos or scars covering more than 50% of the abdominal wall surface area.
22. Participation in other clinical trials and receiving trial interventions within the last 3 months.
23. Existing MRI examination contraindications or inability to cooperate with MRI examinations before screening.
24. Other circumstances deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events (AEs) and Serious Adverse Events | 113 days

SECONDARY OUTCOMES:
The maximum observed serum concentration (Cmax) of B1344. | 113 days
Time to peak serum concentration (Tmax) of B1344 | 113
Area under the serum concentration versus time curve from time zero to the last measurable concentration (AUClast) of B1344 | 113
Terminal elimination half-life (t1/2) of B1344 | 113
Compare the changes in triglycerides (TG) after administration compared to the baseline, as well as the percentage changes. | 90 days
Absolute Change From Baseline in Hepatic Fat Fraction Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) at day 90. | 90 days
Percent Change From Baseline in Hepatic Fat Fraction Assessed by Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI-PDFF) at day 90. | 90 days
The proportion of participants with ≥30% relative fat reduction on MRI-PDFF compared to the baseline at day 90 | 90 days
Absolute Change and Percent Change From Baseline in HbA1c at day 90. | 90 days
The proportion of participants with ≥17U/L reduction on ALT compared to the baseline at day 90. | 90 days
Absolute Change and Percent Change From Baseline in ALT and AST at day 90. | 90 days
Absolute change and percent change from baseline in pro-C3 based on Fibroscan liver stiffness measurement (LSM) at day 90. | 90 days
Absolute Change and Percent Change From Baseline in Body Weight at Day 90. | 90 days

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Tsinghua Changgung Hospital (BTCH) affiliated to Tsinghua University, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sinopharm Tongmei General Hospital, Datong, Shanxi
  - The First Affiliated Hospital to Nankai University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital to Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided